CLINICAL TRIAL: NCT05660824
Title: Effectiveness of Stromal Vascular Fraction (SVF) and Platelet -Rich Plasma (PRP) in Patients With Knee Osteoarthritis: Study Protocol for a Phase III, Prospective, Randomized, Controlled Multi-center Study : (SPOST Study)
Brief Title: Effectiveness of Stromal Vascular Fraction (SVF) and Platelet -Rich Plasma (PRP) in Patients With Knee Osteoarthritis: Study Protocol for a Phase III, Prospective, Randomized, Controlled Multi-center Study.
Acronym: SPOST
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Adrien Schwitzguebel (Other)
Responsible Party: Sponsor-Investigator, Adrien Schwitzguebel, Physician Director of Sports Medicine Department, Hôpital de la Providence, Switzerland
Organization: Hôpital de la Providence, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 28.12.2024
Record Dates: First submitted 2022-01-24; First posted 2022-12-21 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis
Keywords: mesenchymal stem cells; stem cells; Stromal Vascular Fraction; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Multicentric randomized. Randomization will be performed at a 1:1 ratio to either the intervention arm or the active comparator. Each block of 4 patients will be assigned to specific strata according to age (over or under 40), presence of either partial, full cartilage defects or full cartilage defects with bone deformation.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study is triple-blinded concerning (i) the participants during the intervention and throughout the study duration, (ii) the outcome assessor, and (iii) the statistician. The investigator in charge of the injections will be unblinded and therefore will not be assigned to outcomes assessment.
  Follow-up and outcome assessment will be identical for both arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SVF (Stromal vascular fraction) (Experimental): Patients will receive a venepuncture to obtain PRP, and a lipoaspirate to obtain SVF. Then an ultrasonographic guided PRP+SVF injection will be performed.
  Patients will consecutively receive two monthly PRP injections.
  Interventions: Device: Stromal Vascular Fraction infiltration
- PRP (Platelet-rich plasma) (Active Comparator): Patients will receive a venepuncture to obtain PRP, and a sham lipoaspirate. Then an ultrasonographic guided PRP injection will be performed.
  Patients will consecutively receive two monthly PRP injections.
  Interventions: Procedure: Plattelet Rich Plasma infiltration

INTERVENTIONS:
Device: Stromal Vascular Fraction infiltration — Procedure to prepare SVF: In the operations room and after aseptic technic, local anesthesia is applied in the liposuction incision site with lidocaine 1% without epinephrine subcutaneously. 60 ml of tumescent solution are injected. After 15-20 minutes waiting, 15 ml of lipoaspiration per side are recollected into a double syringe. This is centrifuged for 4 minutes at 2.500 rpm and the remaining fat is separated from the other fractions. Two 1.4 mm GEMS syringes are attached together, and fat is transferred at least 30 times from one syringe to the other. Syringe content is again centrifugated for 4 minutes. The oil is discarded and approximately 1.5ml SVF fraction remains.
  Other Names: Autologous conditionned adipose tissue (ACA) kit by Arthrex
  Arms: SVF (Stromal vascular fraction)
Procedure: Plattelet Rich Plasma infiltration — Procedure to prepare PRP: 15 cm of peripheral blood obtained by venipuncture are centrifugated at 1500 RPM during 5 minutes. Using PRP Arthrex kit platelets poor plasma is discarded and 1-3 mm of PRP are ready to be injected
  Other Names: Autologous conditionned plasma (ACP) kit by Arthrex
  Arms: PRP (Platelet-rich plasma)

SUMMARY:
This multicenter, randomized, triple-blind, controlled trial, will enroll 108 patients who will block-randomized in a 1:1 ratio to either the intervention or control group. The main question to answer are the clinical efficacy of SVF as adjuvant therapy to PRP on functionality and tissue regeneration for knee osteoarthritis.

DETAILED DESCRIPTION:
Background:

Osteoarthritis, the most common joint disease, has a high social and individual impact and the development of therapeutic options is a public health priority. It's multifactorial etiology is still a source of active research

Most common conservative treatments for osteoarthritis treatment include painkillers, active physical therapies, orthotics, infiltrations of corticosteroids, hyaluronic acid (HA), and platelet-rich plasma (PRP).

PRP may be beneficial in osteoarthritis by interfering with catabolic and inflammatory events and by subsequently promoting anabolic responses. Activation of PRP releases biologically active components, including platelet-derived growth factor (PDGF), transforming growth factor-β (PGF-β), type I insulin-like growth factor (IGF-1) and vascular endothelial growth factor (VEGF). These proteins are responsible for a range of critical tissue healing roles such as chondrocyte and mesenchymal stem cells proliferation, bone and vessel remodelling, inflammatory modulation and collagen synthesis.

For osteoarthritis, an improvement of clinical outcomes has been found in several clinical trials, presumably associated with the chondroprotective effect of PRP. Nevertheless, an in-vivo effect on human cartilage regeneration is not yet demonstrated despite the numerous studies approaching the subject.

Preclinical models elucidated how injected Adipose Derived- Mesenchymal Stem Cells (AD-MSC) coordinate the cartilage regeneration process through paracrine mechanisms, producing cytokines and trophic bioactive factors that stimulate cellular proliferation, reduce inflammation, fibrosis, oxidative stress, and chondrocytes senescence.

Stromal Vascular Fraction (SVF), a product from specific adipose tissue processing, contains mesenchymal stem cells, endothelial precursor cells, T regulatory cells, macrophages, smooth muscle cells, pericytes and preadipocytes. SVF extraction and injection techniques have been recently used as an alternative to harvest AD-MSC due to its logistic simplicity and feasibility in clinical practice.

SVF injections produce a clinically significant effect on the treatment of knee osteoarthritis, and a possible improvement in cartilage quality.

This clinical trial aims to assess the clinical efficacy of SVF as adjuvant therapy to PRP on functionality and tissue regeneration on osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Age older than 16 years old,
* Symptomatic knee osteoarthritis confirmed by magnetic resonance imaging (MRI)
* Absence of free or displaced meniscal or cartilage fragments on the MRI of the affected knee
* Failure of first-line conservative management in the last 3 months including medical or infiltrative treatment, orthotics use, active rehabilitation plan, adaptation of sports and work habits.

Exclusion Criteria:

* Patient is familiar with the lipoaspiration process
* Significant disease of the contralateral member with a function evaluated with SANE score below 80%
* Microcristalline disease (i.e. gout, pseudogout),
* Active inflammatory rheumatic disorders,
* Need of regular anti-inflammatory treatment (either NSAIDs or corticosteroids),
* Allergy to local anesthetics or epinephrin
* Bleeding disorders or current anticoagulation therapy
* Patients with decompensated renal failure, hepatic dysfunction, or severe pulmonary or cardiovascular disease,
* Patients with an immunocompromised status
* Women who are pregnant or intend to become pregnant during the study
* Inability to follow the procedures of the study, e.g., due to language problems, psychological disorders, dementia, etc. of the participant,
* Known or suspected non-compliance, drug, or alcohol abuse
* Previous enrollment into the current study,
* Participation in another study with investigational drug or procedure within the 30 days preceding and during the present study
* Enrollment of the investigator, his/her family members, employees, and other dependent persons

If a bilateral disease is present and both sides require either the experimental or the control intervention, only the most symptomatic side will be studied.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
WOMAC | 6 months
  Functional improvement measured with the 0%-100% normalized Western Ontario McMaster Universities Osteoarthritis Index, where 0% indicates complete absence of symptoms and 100% indicates maximal possible symptoms severity

SECONDARY OUTCOMES:
VAS | 1, 2, 3, 6, and 12 months
  The absolute difference (changes from baseline to other time points) in pain Visual Analogue Scale (VAS) during maximal physical activity performed by the patient, between the treatment and control arms on a 0 to 10 scale. 0: no pain, 10: maximal pain
WOMAC | 1, 2, 3, 6, and 12 months
  The absolute difference (changes from baseline to other time points) between the treatment and control arms on the Western Ontario McMaster Universities Osteoarthritis Index on knee osteoarthritis cases. From 0 to 100, being 0: no limitation, 100: extreme limitation
Return to work | 1, 2, 3, 6, and 12 months
  The absolute difference between the treatment and control arms on length of time to return work in days
Return to sport | 1, 2, 3, 6, and 12 months
  The absolute difference between the treatment and control arms on length of time to return to sports in days
AMADEUS SCORE | 6 and 12 moths
  The absolute difference (changes from baseline to other time points) between the treatment and control arms on Affected cartilage quality on MRI using Area Measurement And Depth Underlying Structures (AMADEUS) score. (0 worst, 100 best)
WORMS | 6 Months, 12 months
  The absolute difference (changes from baseline to other time points) between the treatment and control arms on Whole-Organ Magnetic Resonance Imaging Score score. (0 normal structure, 332 most severe grade).
MOCART | 6 months, 12 months
  The absolute difference (changes from baseline to other time points) between the treatment and control arms on Magnetic Resonance Observation of Cartilage Repair Tissue score. (0 = poor cartilage repair, 100 complete and normal cartilage repair)

OTHER OUTCOMES:
Age | Baseline
  Age
Sex | Baseline
  Sex
Height | Baseline
  Height, cm
Weight | Baseline
  Weight, kg
BMI | Baseline
  BMI
Number of patients with tobacco use | Baseline
  Number of patients with tobacco use
Number of Participants with concomitant diseases | Baseline
  Number of Participants with concomitant diseases (diabetes Miletus, dyslipidemia, arterial hypertension, osteopenia, osteoporosis, presence of rheumatologic disease, renal failure, and other relevant comorbidity)
Numer of current and previous treatments | Baseline
  Number of current and previous treatments for osteoarthritis and tendinopathy
Kellgren-Lawrence | Baseline
  Baseline Kellgren-Lawrence grade in case of osteoarthritis. I: Mild to IV: Severe
Number of patients with post-traumatic osteoarthritis | Baseline
  Number of patients with post-traumatic osteoarthritis

CONTACTS AND LOCATIONS:
Overall Officials: Adrien Schwitzguébel, MD., Principal Investigator — Hôpital de La Providenc

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Medical A. WMA declaration of Helsinki : ethical principles for medical research involving human subjects 2013. First edition. ed. Guildford, Surrey: Canary Publications; 2014. 12 pages p.
- [Background] Harmonization ICo. Guideline for Good Clinical Practice. 1996.
- [Background] McCormack J, Underwood F, Slaven E, Cappaert T. THE MINIMUM CLINICALLY IMPORTANT DIFFERENCE ON THE VISA-A AND LEFS FOR PATIENTS WITH INSERTIONAL ACHILLES TENDINOPATHY. Int J Sports Phys Ther. 2015 Oct;10(5):639-44. PMID 26491614
- [Background] Franchignoni F, Vercelli S, Giordano A, Sartorio F, Bravini E, Ferriero G. Minimal clinically important difference of the disabilities of the arm, shoulder and hand outcome measure (DASH) and its shortened version (QuickDASH). J Orthop Sports Phys Ther. 2014 Jan;44(1):30-9. doi: 10.2519/jospt.2014.4893. Epub 2013 Oct 30. PMID 24175606
- [Background] Emanuel EJ, Wendler D, Grady C. What makes clinical research ethical? JAMA. 2000 May 24-31;283(20):2701-11. doi: 10.1001/jama.283.20.2701. PMID 10819955
- [Background] Agarwal N, Mak C, Bojanic C, To K, Khan W. Meta-Analysis of Adipose Tissue Derived Cell-Based Therapy for the Treatment of Knee Osteoarthritis. Cells. 2021 Jun 1;10(6):1365. doi: 10.3390/cells10061365. PMID 34206010
- [Background] Ma W, Liu C, Wang S, Xu H, Sun H, Fan X. Efficacy and safety of intra-articular injection of mesenchymal stem cells in the treatment of knee osteoarthritis: A systematic review and meta-analysis. Medicine (Baltimore). 2020 Dec 4;99(49):e23343. doi: 10.1097/MD.0000000000023343. PMID 33285713
- [Background] Zhao D, Pan JK, Yang WY, Han YH, Zeng LF, Liang GH, Liu J. Intra-Articular Injections of Platelet-Rich Plasma, Adipose Mesenchymal Stem Cells, and Bone Marrow Mesenchymal Stem Cells Associated With Better Outcomes Than Hyaluronic Acid and Saline in Knee Osteoarthritis: A Systematic Review and Network Meta-analysis. Arthroscopy. 2021 Jul;37(7):2298-2314.e10. doi: 10.1016/j.arthro.2021.02.045. Epub 2021 Mar 10. PMID 33713757
- [Background] Jiang P, Mao L, Qiao L, Lei X, Zheng Q, Li D. Efficacy and safety of mesenchymal stem cell injections for patients with osteoarthritis: a meta-analysis and review of RCTs. Arch Orthop Trauma Surg. 2021 Jul;141(7):1241-1251. doi: 10.1007/s00402-020-03703-0. Epub 2021 Jan 28. PMID 33507375
- [Background] Dai W, Leng X, Wang J, Shi Z, Cheng J, Hu X, Ao Y. Intra-Articular Mesenchymal Stromal Cell Injections Are No Different From Placebo in the Treatment of Knee Osteoarthritis: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Arthroscopy. 2021 Jan;37(1):340-358. doi: 10.1016/j.arthro.2020.10.016. Epub 2020 Oct 21. PMID 33098949
- [Background] Lee SY, Kim W, Lim C, Chung SG. Treatment of Lateral Epicondylosis by Using Allogeneic Adipose-Derived Mesenchymal Stem Cells: A Pilot Study. Stem Cells. 2015 Oct;33(10):2995-3005. doi: 10.1002/stem.2110. Epub 2015 Aug 6. PMID 26202898
- [Background] Usuelli FG, Grassi M, Maccario C, Vigano' M, Lanfranchi L, Alfieri Montrasio U, de Girolamo L. Intratendinous adipose-derived stromal vascular fraction (SVF) injection provides a safe, efficacious treatment for Achilles tendinopathy: results of a randomized controlled clinical trial at a 6-month follow-up. Knee Surg Sports Traumatol Arthrosc. 2018 Jul;26(7):2000-2010. doi: 10.1007/s00167-017-4479-9. Epub 2017 Mar 1. PMID 28251260
- [Background] Stein BE, Stroh DA, Schon LC. Outcomes of acute Achilles tendon rupture repair with bone marrow aspirate concentrate augmentation. Int Orthop. 2015 May;39(5):901-5. doi: 10.1007/s00264-015-2725-7. Epub 2015 Mar 22. PMID 25795246
- [Background] Kim YS, Sung CH, Chung SH, Kwak SJ, Koh YG. Does an Injection of Adipose-Derived Mesenchymal Stem Cells Loaded in Fibrin Glue Influence Rotator Cuff Repair Outcomes? A Clinical and Magnetic Resonance Imaging Study. Am J Sports Med. 2017 Jul;45(9):2010-2018. doi: 10.1177/0363546517702863. Epub 2017 Apr 27. PMID 28448728
- [Background] Michalek J, Vrablikova A, Darinskas A, Lukac L, Prucha J, Skopalik J, Travnik J, Cibulka M, Dudasova Z. Stromal vascular fraction cell therapy for osteoarthritis in elderly: Multicenter case-control study. J Clin Orthop Trauma. 2019 Jan-Feb;10(1):76-80. doi: 10.1016/j.jcot.2018.11.010. Epub 2018 Nov 23. No abstract available. PMID 30705536
- [Background] Al Faqeh H, Nor Hamdan BM, Chen HC, Aminuddin BS, Ruszymah BH. The potential of intra-articular injection of chondrogenic-induced bone marrow stem cells to retard the progression of osteoarthritis in a sheep model. Exp Gerontol. 2012 Jun;47(6):458-64. doi: 10.1016/j.exger.2012.03.018. Epub 2012 Apr 10. PMID 22759409
- [Background] Awad HA, Boivin GP, Dressler MR, Smith FN, Young RG, Butler DL. Repair of patellar tendon injuries using a cell-collagen composite. J Orthop Res. 2003 May;21(3):420-31. doi: 10.1016/S0736-0266(02)00163-8. PMID 12706014
- [Background] Borakati A, Mafi R, Mafi P, Khan WS. A Systematic Review And Meta-Analysis of Clinical Trials of Mesenchymal Stem Cell Therapy for Cartilage Repair. Curr Stem Cell Res Ther. 2018 Feb 23;13(3):215-225. doi: 10.2174/1574888X12666170915120620. PMID 28914207
- [Background] Chiang ER, Ma HL, Wang JP, Liu CL, Chen TH, Hung SC. Allogeneic Mesenchymal Stem Cells in Combination with Hyaluronic Acid for the Treatment of Osteoarthritis in Rabbits. PLoS One. 2016 Feb 25;11(2):e0149835. doi: 10.1371/journal.pone.0149835. eCollection 2016. PMID 26915044
- [Background] Chong AK, Ang AD, Goh JC, Hui JH, Lim AY, Lee EH, Lim BH. Bone marrow-derived mesenchymal stem cells influence early tendon-healing in a rabbit achilles tendon model. J Bone Joint Surg Am. 2007 Jan;89(1):74-81. doi: 10.2106/JBJS.E.01396. PMID 17200313
- [Background] Comella K, Parlo M, Daly R, Depasquale V, Edgerton E, Mallory P, Schmidt R, Drake WP. Safety Analysis of Autologous Stem Cell Therapy in a Variety of Degenerative Diseases and Injuries Using the Stromal Vascular Fraction. J Clin Med Res. 2017 Nov;9(11):935-942. doi: 10.14740/jocmr3187w. Epub 2017 Oct 2. PMID 29038672
- [Background] Crovace A, Lacitignola L, De Siena R, Rossi G, Francioso E. Cell therapy for tendon repair in horses: an experimental study. Vet Res Commun. 2007 Aug;31 Suppl 1:281-3. doi: 10.1007/s11259-007-0047-y. No abstract available. PMID 17682895
- [Background] Damia E, Chicharro D, Lopez S, Cuervo B, Rubio M, Sopena JJ, Vilar JM, Carrillo JM. Adipose-Derived Mesenchymal Stem Cells: Are They a Good Therapeutic Strategy for Osteoarthritis? Int J Mol Sci. 2018 Jun 30;19(7):1926. doi: 10.3390/ijms19071926. PMID 29966351
- [Background] Davatchi F, Abdollahi BS, Mohyeddin M, Shahram F, Nikbin B. Mesenchymal stem cell therapy for knee osteoarthritis. Preliminary report of four patients. Int J Rheum Dis. 2011 May;14(2):211-5. doi: 10.1111/j.1756-185X.2011.01599.x. Epub 2011 Mar 4. PMID 21518322
- [Background] de Windt TS, Vonk LA, Slaper-Cortenbach ICM, Nizak R, van Rijen MHP, Saris DBF. Allogeneic MSCs and Recycled Autologous Chondrons Mixed in a One-Stage Cartilage Cell Transplantion: A First-in-Man Trial in 35 Patients. Stem Cells. 2017 Aug;35(8):1984-1993. doi: 10.1002/stem.2657. Epub 2017 Jun 23. PMID 28600828
- [Background] Del Bue M, Ricco S, Ramoni R, Conti V, Gnudi G, Grolli S. Equine adipose-tissue derived mesenchymal stem cells and platelet concentrates: their association in vitro and in vivo. Vet Res Commun. 2008 Sep;32 Suppl 1:S51-5. doi: 10.1007/s11259-008-9093-3. PMID 18683070
- [Background] Desando G, Cavallo C, Sartoni F, Martini L, Parrilli A, Veronesi F, Fini M, Giardino R, Facchini A, Grigolo B. Intra-articular delivery of adipose derived stromal cells attenuates osteoarthritis progression in an experimental rabbit model. Arthritis Res Ther. 2013 Jan 29;15(1):R22. doi: 10.1186/ar4156. PMID 23360790
- [Background] Diekman BO, Wu CL, Louer CR, Furman BD, Huebner JL, Kraus VB, Olson SA, Guilak F. Intra-articular delivery of purified mesenchymal stem cells from C57BL/6 or MRL/MpJ superhealer mice prevents posttraumatic arthritis. Cell Transplant. 2013;22(8):1395-408. doi: 10.3727/096368912X653264. Epub 2012 Aug 10. PMID 22889498
- [Background] Doyle EC, Wragg NM, Wilson SL. Intraarticular injection of bone marrow-derived mesenchymal stem cells enhances regeneration in knee osteoarthritis. Knee Surg Sports Traumatol Arthrosc. 2020 Dec;28(12):3827-3842. doi: 10.1007/s00167-020-05859-z. Epub 2020 Jan 31. PMID 32006075
- [Background] Ellera Gomes JL, da Silva RC, Silla LM, Abreu MR, Pellanda R. Conventional rotator cuff repair complemented by the aid of mononuclear autologous stem cells. Knee Surg Sports Traumatol Arthrosc. 2012 Feb;20(2):373-7. doi: 10.1007/s00167-011-1607-9. Epub 2011 Jul 20. PMID 21773831
- [Background] Emadedin M, Aghdami N, Taghiyar L, Fazeli R, Moghadasali R, Jahangir S, Farjad R, Baghaban Eslaminejad M. Intra-articular injection of autologous mesenchymal stem cells in six patients with knee osteoarthritis. Arch Iran Med. 2012 Jul;15(7):422-8. PMID 22724879
- [Background] Emadedin M, Ghorbani Liastani M, Fazeli R, Mohseni F, Moghadasali R, Mardpour S, Hosseini SE, Niknejadi M, Moeininia F, Aghahossein Fanni A, Baghban Eslaminejhad R, Vosough Dizaji A, Labibzadeh N, Mirazimi Bafghi A, Baharvand H, Aghdami N. Long-Term Follow-up of Intra-articular Injection of Autologous Mesenchymal Stem Cells in Patients with Knee, Ankle, or Hip Osteoarthritis. Arch Iran Med. 2015 Jun;18(6):336-44. PMID 26058927
- [Background] Freitag J, Bates D, Wickham J, Shah K, Huguenin L, Tenen A, Paterson K, Boyd R. Adipose-derived mesenchymal stem cell therapy in the treatment of knee osteoarthritis: a randomized controlled trial. Regen Med. 2019 Mar;14(3):213-230. doi: 10.2217/rme-2018-0161. Epub 2019 Feb 14. PMID 30762487
- [Background] Frisbie DD, Kisiday JD, Kawcak CE, Werpy NM, McIlwraith CW. Evaluation of adipose-derived stromal vascular fraction or bone marrow-derived mesenchymal stem cells for treatment of osteoarthritis. J Orthop Res. 2009 Dec;27(12):1675-80. doi: 10.1002/jor.20933. PMID 19544397
- [Background] Gupta PK, Chullikana A, Rengasamy M, Shetty N, Pandey V, Agarwal V, Wagh SY, Vellotare PK, Damodaran D, Viswanathan P, Thej C, Balasubramanian S, Majumdar AS. Efficacy and safety of adult human bone marrow-derived, cultured, pooled, allogeneic mesenchymal stromal cells (Stempeucel(R)): preclinical and clinical trial in osteoarthritis of the knee joint. Arthritis Res Ther. 2016 Dec 20;18(1):301. doi: 10.1186/s13075-016-1195-7. PMID 27993154
- [Background] Han X, Yang B, Zou F, Sun J. Clinical therapeutic efficacy of mesenchymal stem cells derived from adipose or bone marrow for knee osteoarthritis: a meta-analysis of randomized controlled trials. J Comp Eff Res. 2020 Apr;9(5):361-374. doi: 10.2217/cer-2019-0187. Epub 2020 Mar 6. PMID 32141308
- [Background] Hernigou P, Flouzat Lachaniette CH, Delambre J, Zilber S, Duffiet P, Chevallier N, Rouard H. Biologic augmentation of rotator cuff repair with mesenchymal stem cells during arthroscopy improves healing and prevents further tears: a case-controlled study. Int Orthop. 2014 Sep;38(9):1811-8. doi: 10.1007/s00264-014-2391-1. Epub 2014 Jun 7. PMID 24913770
- [Background] Huang R, Li W, Zhao Y, Yang F, Xu M. Clinical efficacy and safety of stem cell therapy for knee osteoarthritis: A meta-analysis. Medicine (Baltimore). 2020 Mar;99(11):e19434. doi: 10.1097/MD.0000000000019434. PMID 32176071
- [Background] Jo CH, Lee YG, Shin WH, Kim H, Chai JW, Jeong EC, Kim JE, Shim H, Shin JS, Shin IS, Ra JC, Oh S, Yoon KS. Intra-articular injection of mesenchymal stem cells for the treatment of osteoarthritis of the knee: a proof-of-concept clinical trial. Stem Cells. 2014 May;32(5):1254-66. doi: 10.1002/stem.1634. PMID 24449146
- [Background] Kalamegam G, Memic A, Budd E, Abbas M, Mobasheri A. A Comprehensive Review of Stem Cells for Cartilage Regeneration in Osteoarthritis. Adv Exp Med Biol. 2018;1089:23-36. doi: 10.1007/5584_2018_205. PMID 29725971
- [Background] Kim SH, Djaja YP, Park YB, Park JG, Ko YB, Ha CW. Intra-articular Injection of Culture-Expanded Mesenchymal Stem Cells Without Adjuvant Surgery in Knee Osteoarthritis: A Systematic Review and Meta-analysis. Am J Sports Med. 2020 Sep;48(11):2839-2849. doi: 10.1177/0363546519892278. Epub 2019 Dec 24. PMID 31874044
- [Background] Kim SH, Ha CW, Park YB, Nam E, Lee JE, Lee HJ. Intra-articular injection of mesenchymal stem cells for clinical outcomes and cartilage repair in osteoarthritis of the knee: a meta-analysis of randomized controlled trials. Arch Orthop Trauma Surg. 2019 Jul;139(7):971-980. doi: 10.1007/s00402-019-03140-8. Epub 2019 Feb 11. PMID 30756165
- [Background] Kim YS, Choi YJ, Lee SW, Kwon OR, Suh DS, Heo DB, Koh YG. Assessment of clinical and MRI outcomes after mesenchymal stem cell implantation in patients with knee osteoarthritis: a prospective study. Osteoarthritis Cartilage. 2016 Feb;24(2):237-45. doi: 10.1016/j.joca.2015.08.009. Epub 2015 Aug 28. PMID 26318655
- [Background] Kim YS, Choi YJ, Suh DS, Heo DB, Kim YI, Ryu JS, Koh YG. Mesenchymal stem cell implantation in osteoarthritic knees: is fibrin glue effective as a scaffold? Am J Sports Med. 2015 Jan;43(1):176-85. doi: 10.1177/0363546514554190. Epub 2014 Oct 27. PMID 25349263
- [Background] Kim YS, Koh YG. Injection of Mesenchymal Stem Cells as a Supplementary Strategy of Marrow Stimulation Improves Cartilage Regeneration After Lateral Sliding Calcaneal Osteotomy for Varus Ankle Osteoarthritis: Clinical and Second-Look Arthroscopic Results. Arthroscopy. 2016 May;32(5):878-89. doi: 10.1016/j.arthro.2016.01.020. Epub 2016 Mar 15. PMID 26993668
- [Background] Kim YS, Kwon OR, Choi YJ, Suh DS, Heo DB, Koh YG. Comparative Matched-Pair Analysis of the Injection Versus Implantation of Mesenchymal Stem Cells for Knee Osteoarthritis. Am J Sports Med. 2015 Nov;43(11):2738-46. doi: 10.1177/0363546515599632. Epub 2015 Sep 3. PMID 26337418
- [Background] Kim YS, Lee M, Koh YG. Additional mesenchymal stem cell injection improves the outcomes of marrow stimulation combined with supramalleolar osteotomy in varus ankle osteoarthritis: short-term clinical results with second-look arthroscopic evaluation. J Exp Orthop. 2016 Dec;3(1):12. doi: 10.1186/s40634-016-0048-2. Epub 2016 May 20. PMID 27206975
- [Background] Koh YG, Choi YJ. Infrapatellar fat pad-derived mesenchymal stem cell therapy for knee osteoarthritis. Knee. 2012 Dec;19(6):902-7. doi: 10.1016/j.knee.2012.04.001. Epub 2012 May 14. PMID 22583627
- [Background] Koh YG, Kwon OR, Kim YS, Choi YJ. Comparative outcomes of open-wedge high tibial osteotomy with platelet-rich plasma alone or in combination with mesenchymal stem cell treatment: a prospective study. Arthroscopy. 2014 Nov;30(11):1453-60. doi: 10.1016/j.arthro.2014.05.036. Epub 2014 Aug 6. PMID 25108907
- [Background] Lacitignola L, Crovace A, Rossi G, Francioso E. Cell therapy for tendinitis, experimental and clinical report. Vet Res Commun. 2008 Sep;32 Suppl 1:S33-8. doi: 10.1007/s11259-008-9085-3. PMID 18686004
- [Background] Lamo-Espinosa JM, Mora G, Blanco JF, Granero-Molto F, Nunez-Cordoba JM, Lopez-Elio S, Andreu E, Sanchez-Guijo F, Aquerreta JD, Bondia JM, Valenti-Azcarate A, Del Consuelo Del Canizo M, Villaron EM, Valenti-Nin JR, Prosper F. Intra-articular injection of two different doses of autologous bone marrow mesenchymal stem cells versus hyaluronic acid in the treatment of knee osteoarthritis: long-term follow up of a multicenter randomized controlled clinical trial (phase I/II). J Transl Med. 2018 Jul 31;16(1):213. doi: 10.1186/s12967-018-1591-7. PMID 30064455
- [Background] Lee JM, Im GI. SOX trio-co-transduced adipose stem cells in fibrin gel to enhance cartilage repair and delay the progression of osteoarthritis in the rat. Biomaterials. 2012 Mar;33(7):2016-24. doi: 10.1016/j.biomaterials.2011.11.050. Epub 2011 Dec 19. PMID 22189147
- [Background] Lee KB, Hui JH, Song IC, Ardany L, Lee EH. Injectable mesenchymal stem cell therapy for large cartilage defects--a porcine model. Stem Cells. 2007 Nov;25(11):2964-71. doi: 10.1634/stemcells.2006-0311. Epub 2007 Jul 26. PMID 17656639
- [Background] Lee WS, Kim HJ, Kim KI, Kim GB, Jin W. Intra-Articular Injection of Autologous Adipose Tissue-Derived Mesenchymal Stem Cells for the Treatment of Knee Osteoarthritis: A Phase IIb, Randomized, Placebo-Controlled Clinical Trial. Stem Cells Transl Med. 2019 Jun;8(6):504-511. doi: 10.1002/sctm.18-0122. Epub 2019 Mar 5. PMID 30835956
- [Background] Lu L, Dai C, Du H, Li S, Ye P, Zhang L, Wang X, Song Y, Togashi R, Vangsness CT, Bao C. Intra-articular injections of allogeneic human adipose-derived mesenchymal progenitor cells in patients with symptomatic bilateral knee osteoarthritis: a Phase I pilot study. Regen Med. 2020 May;15(5):1625-1636. doi: 10.2217/rme-2019-0106. Epub 2020 Jul 17. PMID 32677876
- [Background] Lu L, Dai C, Zhang Z, Du H, Li S, Ye P, Fu Q, Zhang L, Wu X, Dong Y, Song Y, Zhao D, Pang Y, Bao C. Treatment of knee osteoarthritis with intra-articular injection of autologous adipose-derived mesenchymal progenitor cells: a prospective, randomized, double-blind, active-controlled, phase IIb clinical trial. Stem Cell Res Ther. 2019 May 21;10(1):143. doi: 10.1186/s13287-019-1248-3. PMID 31113476
- [Background] Maheshwer B, Polce EM, Paul K, Williams BT, Wolfson TS, Yanke A, Verma NN, Cole BJ, Chahla J. Regenerative Potential of Mesenchymal Stem Cells for the Treatment of Knee Osteoarthritis and Chondral Defects: A Systematic Review and Meta-analysis. Arthroscopy. 2021 Jan;37(1):362-378. doi: 10.1016/j.arthro.2020.05.037. Epub 2020 Jun 1. PMID 32497658
- [Background] Mianehsaz E, Mirzaei HR, Mahjoubin-Tehran M, Rezaee A, Sahebnasagh R, Pourhanifeh MH, Mirzaei H, Hamblin MR. Mesenchymal stem cell-derived exosomes: a new therapeutic approach to osteoarthritis? Stem Cell Res Ther. 2019 Nov 21;10(1):340. doi: 10.1186/s13287-019-1445-0. PMID 31753036
- [Background] Mizuno K, Muneta T, Morito T, Ichinose S, Koga H, Nimura A, Mochizuki T, Sekiya I. Exogenous synovial stem cells adhere to defect of meniscus and differentiate into cartilage cells. J Med Dent Sci. 2008 Mar;55(1):101-11. PMID 19845155
- [Background] Muhammad SA, Nordin N, Mehat MZ, Fakurazi S. Comparative efficacy of stem cells and secretome in articular cartilage regeneration: a systematic review and meta-analysis. Cell Tissue Res. 2019 Feb;375(2):329-344. doi: 10.1007/s00441-018-2884-0. Epub 2018 Aug 6. PMID 30084022
- [Background] Murphy JM, Fink DJ, Hunziker EB, Barry FP. Stem cell therapy in a caprine model of osteoarthritis. Arthritis Rheum. 2003 Dec;48(12):3464-74. doi: 10.1002/art.11365. PMID 14673997
- [Background] Orozco L, Munar A, Soler R, Alberca M, Soler F, Huguet M, Sentis J, Sanchez A, Garcia-Sancho J. Treatment of knee osteoarthritis with autologous mesenchymal stem cells: a pilot study. Transplantation. 2013 Jun 27;95(12):1535-41. doi: 10.1097/TP.0b013e318291a2da. PMID 23680930
- [Background] Ouyang HW, Goh JC, Thambyah A, Teoh SH, Lee EH. Knitted poly-lactide-co-glycolide scaffold loaded with bone marrow stromal cells in repair and regeneration of rabbit Achilles tendon. Tissue Eng. 2003 Jun;9(3):431-9. doi: 10.1089/107632703322066615. PMID 12857411
- [Background] Park YB, Ha CW, Kim JA, Han WJ, Rhim JH, Lee HJ, Kim KJ, Park YG, Chung JY. Single-stage cell-based cartilage repair in a rabbit model: cell tracking and in vivo chondrogenesis of human umbilical cord blood-derived mesenchymal stem cells and hyaluronic acid hydrogel composite. Osteoarthritis Cartilage. 2017 Apr;25(4):570-580. doi: 10.1016/j.joca.2016.10.012. Epub 2016 Oct 24. PMID 27789339
- [Background] Pascual-Garrido C, Rolon A, Makino A. Treatment of chronic patellar tendinopathy with autologous bone marrow stem cells: a 5-year-followup. Stem Cells Int. 2012;2012:953510. doi: 10.1155/2012/953510. Epub 2011 Dec 18. PMID 22220180
- [Background] Ruster B, Gottig S, Ludwig RJ, Bistrian R, Muller S, Seifried E, Gille J, Henschler R. Mesenchymal stem cells display coordinated rolling and adhesion behavior on endothelial cells. Blood. 2006 Dec 1;108(12):3938-44. doi: 10.1182/blood-2006-05-025098. Epub 2006 Aug 8. PMID 16896152
- [Background] Shariatzadeh M, Song J, Wilson SL. The efficacy of different sources of mesenchymal stem cells for the treatment of knee osteoarthritis. Cell Tissue Res. 2019 Dec;378(3):399-410. doi: 10.1007/s00441-019-03069-9. Epub 2019 Jul 15. PMID 31309317
- [Background] Smith RK, Webbon PM. Harnessing the stem cell for the treatment of tendon injuries: heralding a new dawn? Br J Sports Med. 2005 Sep;39(9):582-4. doi: 10.1136/bjsm.2005.015834. No abstract available. PMID 16118291
- [Background] Song Y, Du H, Dai C, Zhang L, Li S, Hunter DJ, Lu L, Bao C. Human adipose-derived mesenchymal stem cells for osteoarthritis: a pilot study with long-term follow-up and repeated injections. Regen Med. 2018 Apr;13(3):295-307. doi: 10.2217/rme-2017-0152. Epub 2018 Feb 8. PMID 29417902
- [Background] Spasovski D, Spasovski V, Bascarevic Z, Stojiljkovic M, Vreca M, Andelkovic M, Pavlovic S. Intra-articular injection of autologous adipose-derived mesenchymal stem cells in the treatment of knee osteoarthritis. J Gene Med. 2018 Jan;20(1). doi: 10.1002/jgm.3002. Epub 2018 Jan 22. PMID 29243283
- [Background] Steingen C, Brenig F, Baumgartner L, Schmidt J, Schmidt A, Bloch W. Characterization of key mechanisms in transmigration and invasion of mesenchymal stem cells. J Mol Cell Cardiol. 2008 Jun;44(6):1072-1084. doi: 10.1016/j.yjmcc.2008.03.010. Epub 2008 Mar 19. PMID 18462748
- [Background] Suhaeb AM, Naveen S, Mansor A, Kamarul T. Hyaluronic acid with or without bone marrow derived-mesenchymal stem cells improves osteoarthritic knee changes in rat model: a preliminary report. Indian J Exp Biol. 2012 Jun;50(6):383-90. PMID 22734248
- [Background] ter Huurne M, Schelbergen R, Blattes R, Blom A, de Munter W, Grevers LC, Jeanson J, Noel D, Casteilla L, Jorgensen C, van den Berg W, van Lent PL. Antiinflammatory and chondroprotective effects of intraarticular injection of adipose-derived stem cells in experimental osteoarthritis. Arthritis Rheum. 2012 Nov;64(11):3604-13. doi: 10.1002/art.34626. PMID 22961401
- [Background] Toghraie F, Razmkhah M, Gholipour MA, Faghih Z, Chenari N, Torabi Nezhad S, Nazhvani Dehghani S, Ghaderi A. Scaffold-free adipose-derived stem cells (ASCs) improve experimentally induced osteoarthritis in rabbits. Arch Iran Med. 2012 Aug;15(8):495-9. PMID 22827787
- [Background] Toghraie FS, Chenari N, Gholipour MA, Faghih Z, Torabinejad S, Dehghani S, Ghaderi A. Treatment of osteoarthritis with infrapatellar fat pad derived mesenchymal stem cells in Rabbit. Knee. 2011 Mar;18(2):71-5. doi: 10.1016/j.knee.2010.03.001. Epub 2010 Jun 29. PMID 20591677
- [Background] Ude CC, Sulaiman SB, Min-Hwei N, Hui-Cheng C, Ahmad J, Yahaya NM, Saim AB, Idrus RB. Cartilage regeneration by chondrogenic induced adult stem cells in osteoarthritic sheep model. PLoS One. 2014 Jun 9;9(6):e98770. doi: 10.1371/journal.pone.0098770. eCollection 2014. PMID 24911365
- [Background] Van Pham P, Hong-Thien Bui K, Quoc Ngo D, Tan Khuat L, Kim Phan N. Transplantation of Nonexpanded Adipose Stromal Vascular Fraction and Platelet-Rich Plasma for Articular Cartilage Injury Treatment in Mice Model. J Med Eng. 2013;2013:832396. doi: 10.1155/2013/832396. Epub 2013 Jan 16. PMID 27006923
- [Background] Vangsness CT Jr, Farr J 2nd, Boyd J, Dellaero DT, Mills CR, LeRoux-Williams M. Adult human mesenchymal stem cells delivered via intra-articular injection to the knee following partial medial meniscectomy: a randomized, double-blind, controlled study. J Bone Joint Surg Am. 2014 Jan 15;96(2):90-8. doi: 10.2106/JBJS.M.00058. PMID 24430407
- [Background] Vega A, Martin-Ferrero MA, Del Canto F, Alberca M, Garcia V, Munar A, Orozco L, Soler R, Fuertes JJ, Huguet M, Sanchez A, Garcia-Sancho J. Treatment of Knee Osteoarthritis With Allogeneic Bone Marrow Mesenchymal Stem Cells: A Randomized Controlled Trial. Transplantation. 2015 Aug;99(8):1681-90. doi: 10.1097/TP.0000000000000678. PMID 25822648
- [Background] Wakitani S, Imoto K, Yamamoto T, Saito M, Murata N, Yoneda M. Human autologous culture expanded bone marrow mesenchymal cell transplantation for repair of cartilage defects in osteoarthritic knees. Osteoarthritis Cartilage. 2002 Mar;10(3):199-206. doi: 10.1053/joca.2001.0504. PMID 11869080
- [Background] Wang J, Guo X, Kang Z, Qi L, Yang Y, Wang J, Xu J, Gao S. Roles of Exosomes from Mesenchymal Stem Cells in Treating Osteoarthritis. Cell Reprogram. 2020 Jun;22(3):107-117. doi: 10.1089/cell.2019.0098. Epub 2020 May 4. PMID 32364765
- [Background] Wong KL, Lee KB, Tai BC, Law P, Lee EH, Hui JH. Injectable cultured bone marrow-derived mesenchymal stem cells in varus knees with cartilage defects undergoing high tibial osteotomy: a prospective, randomized controlled clinical trial with 2 years' follow-up. Arthroscopy. 2013 Dec;29(12):2020-8. doi: 10.1016/j.arthro.2013.09.074. PMID 24286801
- [Background] Xia P, Wang X, Lin Q, Li X. Efficacy of mesenchymal stem cells injection for the management of knee osteoarthritis: a systematic review and meta-analysis. Int Orthop. 2015 Dec;39(12):2363-72. doi: 10.1007/s00264-015-2785-8. Epub 2015 May 6. PMID 25944079
- [Background] Zhou W, Lin J, Zhao K, Jin K, He Q, Hu Y, Feng G, Cai Y, Xia C, Liu H, Shen W, Hu X, Ouyang H. Single-Cell Profiles and Clinically Useful Properties of Human Mesenchymal Stem Cells of Adipose and Bone Marrow Origin. Am J Sports Med. 2019 Jun;47(7):1722-1733. doi: 10.1177/0363546519848678. Epub 2019 May 17. PMID 31100005
- [Background] Zwolanek D, Satue M, Proell V, Godoy JR, Odorfer KI, Flicker M, Hoffmann SC, Rulicke T, Erben RG. Tracking mesenchymal stem cell contributions to regeneration in an immunocompetent cartilage regeneration model. JCI Insight. 2017 Oct 19;2(20):e87322. doi: 10.1172/jci.insight.87322. PMID 29046476
- [Background] Cieza A, Causey K, Kamenov K, Hanson SW, Chatterji S, Vos T. Global estimates of the need for rehabilitation based on the Global Burden of Disease study 2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2021 Dec 19;396(10267):2006-2017. doi: 10.1016/S0140-6736(20)32340-0. Epub 2020 Dec 1. PMID 33275908
- [Background] Musumeci G, Aiello FC, Szychlinska MA, Di Rosa M, Castrogiovanni P, Mobasheri A. Osteoarthritis in the XXIst century: risk factors and behaviours that influence disease onset and progression. Int J Mol Sci. 2015 Mar 16;16(3):6093-112. doi: 10.3390/ijms16036093. PMID 25785564
- [Background] Skjong CC, Meininger AK, Ho SS. Tendinopathy treatment: where is the evidence? Clin Sports Med. 2012 Apr;31(2):329-50. doi: 10.1016/j.csm.2011.11.003. PMID 22341021
- [Background] Chappell AS, Desaiah D, Liu-Seifert H, Zhang S, Skljarevski V, Belenkov Y, Brown JP. A double-blind, randomized, placebo-controlled study of the efficacy and safety of duloxetine for the treatment of chronic pain due to osteoarthritis of the knee. Pain Pract. 2011 Jan-Feb;11(1):33-41. doi: 10.1111/j.1533-2500.2010.00401.x. PMID 20602715
- [Background] Zhang W, Ouyang H, Dass CR, Xu J. Current research on pharmacologic and regenerative therapies for osteoarthritis. Bone Res. 2016 Mar 1;4:15040. doi: 10.1038/boneres.2015.40. eCollection 2016. PMID 26962464
- [Background] Boffa A, Previtali D, Di Laura Frattura G, Vannini F, Candrian C, Filardo G. Evidence on ankle injections for osteochondral lesions and osteoarthritis: a systematic review and meta-analysis. Int Orthop. 2021 Feb;45(2):509-523. doi: 10.1007/s00264-020-04689-5. Epub 2020 Jul 9. PMID 32647968
- [Background] Rees JD, Wolman RL, Wilson A. Eccentric exercises; why do they work, what are the problems and how can we improve them? Br J Sports Med. 2009 Apr;43(4):242-6. doi: 10.1136/bjsm.2008.052910. Epub 2008 Nov 3. PMID 18981040
- [Background] Wilson JJ, Best TM. Common overuse tendon problems: A review and recommendations for treatment. Am Fam Physician. 2005 Sep 1;72(5):811-8. PMID 16156339
- [Background] McCallum SD, Paoloni JA, Murrell GA. Five-year prospective comparison study of topical glyceryl trinitrate treatment of chronic lateral epicondylosis at the elbow. Br J Sports Med. 2011 Apr;45(5):416-20. doi: 10.1136/bjsm.2009.061002. Epub 2009 Jun 23. PMID 19553221
- [Background] Kane SF, Olewinski LH, Tamminga KS. Management of Chronic Tendon Injuries. Am Fam Physician. 2019 Aug 1;100(3):147-157. PMID 31361101
- [Background] Coombes BK, Bisset L, Vicenzino B. Efficacy and safety of corticosteroid injections and other injections for management of tendinopathy: a systematic review of randomised controlled trials. Lancet. 2010 Nov 20;376(9754):1751-67. doi: 10.1016/S0140-6736(10)61160-9. Epub 2010 Oct 21. PMID 20970844
- [Background] Dean BJ, Lostis E, Oakley T, Rombach I, Morrey ME, Carr AJ. The risks and benefits of glucocorticoid treatment for tendinopathy: a systematic review of the effects of local glucocorticoid on tendon. Semin Arthritis Rheum. 2014 Feb;43(4):570-6. doi: 10.1016/j.semarthrit.2013.08.006. Epub 2013 Sep 26. PMID 24074644
- [Background] Wiggins ME, Fadale PD, Ehrlich MG, Walsh WR. Effects of local injection of corticosteroids on the healing of ligaments. A follow-up report. J Bone Joint Surg Am. 1995 Nov;77(11):1682-91. doi: 10.2106/00004623-199511000-00006. PMID 7593077
- [Background] Moraes VY, Lenza M, Tamaoki MJ, Faloppa F, Belloti JC. Platelet-rich therapies for musculoskeletal soft tissue injuries. Cochrane Database Syst Rev. 2013 Dec 23;(12):CD010071. doi: 10.1002/14651858.CD010071.pub2. PMID 24363098
- [Background] Franchini M, Cruciani M, Mengoli C, Marano G, Pupella S, Veropalumbo E, Masiello F, Pati I, Vaglio S, Liumbruno GM. Efficacy of platelet-rich plasma as conservative treatment in orthopaedics: a systematic review and meta-analysis. Blood Transfus. 2018 Nov;16(6):502-513. doi: 10.2450/2018.0111-18. Epub 2018 Sep 3. PMID 30201082
- [Background] Fitzpatrick J, Bulsara M, Zheng MH. The Effectiveness of Platelet-Rich Plasma in the Treatment of Tendinopathy: A Meta-analysis of Randomized Controlled Clinical Trials. Am J Sports Med. 2017 Jan;45(1):226-233. doi: 10.1177/0363546516643716. Epub 2016 Jul 21. PMID 27268111
- [Background] Krogh TP, Ellingsen T, Christensen R, Jensen P, Fredberg U. Ultrasound-Guided Injection Therapy of Achilles Tendinopathy With Platelet-Rich Plasma or Saline: A Randomized, Blinded, Placebo-Controlled Trial. Am J Sports Med. 2016 Aug;44(8):1990-7. doi: 10.1177/0363546516647958. Epub 2016 Jun 2. PMID 27257167
- [Background] Jacobson JA, Yablon CM, Henning PT, Kazmers IS, Urquhart A, Hallstrom B, Bedi A, Parameswaran A. Greater Trochanteric Pain Syndrome: Percutaneous Tendon Fenestration Versus Platelet-Rich Plasma Injection for Treatment of Gluteal Tendinosis. J Ultrasound Med. 2016 Nov;35(11):2413-2420. doi: 10.7863/ultra.15.11046. Epub 2016 Sep 23. PMID 27663654
- [Background] Woodley BL, Newsham-West RJ, Baxter GD. Chronic tendinopathy: effectiveness of eccentric exercise. Br J Sports Med. 2007 Apr;41(4):188-98; discussion 199. doi: 10.1136/bjsm.2006.029769. Epub 2006 Oct 24. PMID 17062655
- [Background] Speed C. A systematic review of shockwave therapies in soft tissue conditions: focusing on the evidence. Br J Sports Med. 2014 Nov;48(21):1538-42. doi: 10.1136/bjsports-2012-091961. Epub 2013 Aug 5. PMID 23918444
- [Background] Zheng C, Zeng D, Chen J, Liu S, Li J, Ruan Z, Liang W. Effectiveness of extracorporeal shock wave therapy in patients with tennis elbow: A meta-analysis of randomized controlled trials. Medicine (Baltimore). 2020 Jul 24;99(30):e21189. doi: 10.1097/MD.0000000000021189. PMID 32791694
- [Background] Mani-Babu S, Morrissey D, Waugh C, Screen H, Barton C. The effectiveness of extracorporeal shock wave therapy in lower limb tendinopathy: a systematic review. Am J Sports Med. 2015 Mar;43(3):752-61. doi: 10.1177/0363546514531911. Epub 2014 May 9. PMID 24817008
- [Background] Maumus M, Pers YM, Ruiz M, Jorgensen C, Noel D. [Mesenchymal stem cells and regenerative medicine: future perspectives in osteoarthritis]. Med Sci (Paris). 2018 Dec;34(12):1092-1099. doi: 10.1051/medsci/2018294. Epub 2019 Jan 9. French. PMID 30623767
- [Background] McGonagle D, Baboolal TG, Jones E. Native joint-resident mesenchymal stem cells for cartilage repair in osteoarthritis. Nat Rev Rheumatol. 2017 Dec;13(12):719-730. doi: 10.1038/nrrheum.2017.182. Epub 2017 Nov 9. PMID 29118440
- [Background] Nguyen A, Guo J, Banyard DA, Fadavi D, Toranto JD, Wirth GA, Paydar KZ, Evans GR, Widgerow AD. Stromal vascular fraction: A regenerative reality? Part 1: Current concepts and review of the literature. J Plast Reconstr Aesthet Surg. 2016 Feb;69(2):170-9. doi: 10.1016/j.bjps.2015.10.015. Epub 2015 Oct 31. PMID 26565755
- [Background] You D, Jang MJ, Kim BH, Song G, Lee C, Suh N, Jeong IG, Ahn TY, Kim CS. Comparative study of autologous stromal vascular fraction and adipose-derived stem cells for erectile function recovery in a rat model of cavernous nerve injury. Stem Cells Transl Med. 2015 Apr;4(4):351-8. doi: 10.5966/sctm.2014-0161. PMID 25792486
- [Background] 112. U.S. DOHAHS. Common Terminology Criteria for Adverse Events (CTCAE) v5.0. November 27, 2017 ed2017.
- [Derived] Schwitzguebel A, Ramirez Cadavid DA, Da Silva T, Decavel P, Benaim C. Effectiveness of Stromal Vascular Fraction (SVF) and Platelet-Rich Plasma (PRP) in Patients With Knee Osteoarthritis: Protocol for a Phase 3, Prospective, Randomized, Controlled, Multicenter Study (SPOST Study). JMIR Res Protoc. 2025 Apr 8;14:e62659. doi: 10.2196/62659. PMID 40198111